CLINICAL TRIAL: NCT02922452
Title: An Open-Label, Single-Sequence Study to Evaluate the Effect of Diltiazem on the Single-Dose Pharmacokinetics of BMS-986141 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Diltiazem on the Pharmacokinetics (PK) of BMS-986141 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV006-028
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — BMS-986141

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-986141 and Dilitazem (Experimental)
  Interventions: Drug: BMS-986141; Drug: Dilitazem

INTERVENTIONS:
Drug: BMS-986141 — Single dose BMS-986141 and Multiple doses of Dilitazem
Drug: Dilitazem — Single dose BMS-986141 and Multiple doses of Dilitazem

SUMMARY:
This study is to evaluate the effect of dilitazem on the single-dose PK of BMS-986141 with parameters like Cmax, AUC(INF), and AUC(0-T).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Healthy men and women (not of child bearing potential) as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests including coagulation parameters.
3. Subjects with body mass index of 18 to 32 kg/m2, inclusive.
4. Women participants must have documented proof that they are not of childbearing potential.
5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-986141 plus 5 half-lives plus 90 days for a total of 100 days post-treatment completion.

Exclusion Criteria:

1. Acute or chronic medical illness, subjects with bleeding diathesis, gastrointestinal ulcer, hepatic disease.
2. History of nausea, diarrhoea, recent surgery, use of tobacco or nicotine containing products, drug or alcohol use, important arrhythmias, sinus bradycardia, chronic headaches, history of multiple events of dizziness, periodontal disease and recent blood donation.
3. Prior exposure to BMS-986141 or prothrombin complex, any investigational product or placebo within 4 weeks of study treatment start, any prescription or over the counter drugs except those cleared by BMS clinical monitor.
4. History of allergy to BMS-986141, dilitazem or any other significant drug allergy or adverse reaction to anticoagulants or antiplatelets.
5. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations beyond what is consistent with the target population

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Days 1-21
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Days 1-21
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC (0-T)) | Days 1-21

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Screening- until 30 days after discontinuation of dosing or subject's participation in the study if the last]

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx